CLINICAL TRIAL: NCT04922567
Title: Multi-center Randomized Study to Compare Efficacy and Safety of Lenalidomide Plus CHOP (L-CHOP) Versus CHOP in Patients With Previously Untreated Peripheral T-cell Lymphoma
Brief Title: Efficacy and Safety of Lenalidomide Plus CHOP vs CHOP in Patients With Untreated Peripheral T-Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Ruijin Hospital (Other); Xinqiao Hospital of Chongqing (Other); Union hospital of Fujian Medical University (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Southern Medical University, China (Other); Shandong Provincial Hospital (Other Government); Huashan Hospital (Other); First Hospital of China Medical University (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Henan Provincial People's Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Changhai Hospital (Other); The Affiliated Hospital of Xuzhou Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); RenJi Hospital (Other); Zhongda Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); Hunan Cancer Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); Xiangya Hospital of Central South University (Other); The First Affiliated Hospital of Dalian Medical University (Other); Jilin Provincial Tumor Hospital (Other); Shanxi Province Cancer Hospital (Other); Zhongshan Hospital Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR2020002513
Record Dates: First submitted 2021-06-05; First posted 2021-06-10 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-10

CONDITIONS: Peripheral T-Cell Lymphoma; Lenalidomide; CHOP
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Lenalidomide; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lenalidomide + CHOP regimen (Experimental)
  Interventions: Drug: Lenalidomide; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone
- CHOP regimen (Active Comparator)
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Lenalidomide — 25mg po on day 1-10
  Arms: lenalidomide + CHOP regimen
Drug: Cyclophosphamide — 750mg/m² iv on day1
Drug: Doxorubicin — 50mg/m² iv on day 1
Drug: Vincristine — 1.4mg/m² iv on day 1
Drug: Prednisone — 100mg po on day1-5

SUMMARY:
This study aims to compare the efficacy and safety of lenalidomide plus CHOP (L-CHOP) versus CHOP alone in patients with previously untreated peripheral T-cell lymphoma (PTCL)

DETAILED DESCRIPTION:
This is a randomized, multi-center, open-label study to compare efficacy and safety of L-CHOP with standard CHOP regimen in patients with previously untreated PTCL. Study subjects are patients with histologically proven PTCL. Patients are randomized 1:1 to receive either cyclophosphamide, doxorubicin, vincristine and prednisone (CHOP) administered in 3 week cycles for 6 cycles or Lenalidomide plus CHOP (L-CHOP) administered in 3 week cycles for 6 cycles. In the L-CHOP arm, Lenalidomide will be administered at a dose of 25mg po on day 1-10 every 3 weeks. This study is divided into three phases: screening phase, treatment phase and follow-up phase. Patients will receive study drug(s) for up to 6 cycles, or until unacceptable toxicity will develop or progression or voluntary with drawl. Adverse event of every treatment cycle will be recorded. Therapy efficacy will be evaluated after finishing 3 cycles and finishing 6 cycles therapy. Patients will be followed until disease progression, died or 3 years from the last patient randomized.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven untreated peripheral T-cell lymphoma (include PTCL not otherwise specified, angioimmunoblastic T cell lymphoma, anaplastic large cell lymphoma, enteropathy-associated T cell lymphoma, Monomorphic epitheliotropic intestinal T-cell lymphoma, Nodal peripheral T-cell lymphoma with T-follicular helper phenotype and Follicular T-cell lymphoma).
2. Males and females of 18 years of age to 80 years of age.
3. Patients have not received anti-tumor therapy.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2.
5. Fit chemotherapy indications and basic requirements, including no obvious abnormal function of heart, liver, lung and kidney: creatine ≤2.0×ULN, total bilirubin ≤2.0mg/dl, transaminases≤3×ULN.
6. Normal peripheral hemogram: absolute neutrophil count(ANC)≥1.5×10^9/L, hemoglobin(Hb)≥90g/L, platelet(PLT)≥100×10^12/L.
7. None of other serious disease conflict with the therapeutic regimen.
8. None of other malignant tumor.
9. Pregnancy test of women at reproductive age must be negative.
10. Estimated survival time ≥ 3 months with good compliance.
11. Voluntary participation, cooperate with the experimental observation, and sign a written informed consent.

Exclusion Criteria:

1. Patients with the following PTCL subtypes are excluded; extranodal natural killer(NK)/T-cell lymphoma, T-prolymphocytic leukemia, T large granular lymphocytic leukemia, chronic lymphoproliferative disorder of NK cells, aggressive NK-cell leukemia, adult T-cell leukemia/ lymphoma, hepatosplenic T-cell lymphoma, subcutaneous panniculitis-like T-cell lymphoma, cutaneous T cell lymphoma, breast implant-associated anaplastic large-cell lymphoma.
2. Transformed lymphoma.
3. Patients with other malignancies in the past or now; or secondary lymphoma triggered by chemotherapy or radiotherapy of other malignancies.
4. Already initiated lymphoma therapy (except for the prephase treatment specified for this study).
5. Patients with primary central nervous system lymphoma or lymphoma involving central nervous system.
6. Patients who have central nervous system or meninges involvements.
7. Candidate for hematopoietic stem cell transplantation.
8. Known hypersensitivity to medications to be used.
9. Hemogram abnormality: ANC<1.5×10^9/L; or hemoglobin<90 g/L; or PLT<100×10^9/L.
10. Known hepatic and renal insufficiency (creatine>2.0×ULN, total bilirubin>2.0 mg/dl，transaminases>3.0×ULN).
11. Patients with decompensated heart failure; or with dilated cardiomyopathy; or with coronary heart disease of non-corresponding ST-segment in ECG diagnosis; or with myocardial infarction within 6 months.
12. Patients with serious uncontrolled acute infection need to be treated with antibody therapies, or antiviral therapies; or serious accompanying disorder or impaired organ function.
13. Know HIV-positivity; or HbsAg positivity; or hepatitis C virus-Ab positivity.
14. Pregnancy or lactation period.
15. Patients who participated in other clinical trials within 3 months.
16. The researchers considered that patients should not be in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response rate | At the end of Cycle 6 (each cycle is 21 days)
  complete response (CR) and partial response (PR) rates, using the standard response criteria( 2014 Lugano criteria)

SECONDARY OUTCOMES:
Progression Free Survival | 3 years
  from date of inclusion to date of progression, relapse, or death from any cause
Overall Survival | 3 years
  From the date of inclusion to date of death, irrespective of cause
Adverse Events | 3 years
  Any unfavorable and unintended sign , symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No